CLINICAL TRIAL: NCT00207701
Title: A Randomized, Double-blind Trial of the Efficacy of REMICADE (Infliximab) Compared With Placebo in Subjects With Ankylosing Spondylitis Receiving Standard Anti-inflammatory Drug Therapy
Brief Title: A Study of Infliximab (Remicade) in Patients With Ankylosing Spondylitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004792; NCT01128504 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; infusion
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab

SUMMARY:
A study of the safety and efficacy of Infliximab (Remicade) versus placebo in subjects with Ankylosing Spondylitis

DETAILED DESCRIPTION:
This is a clinical research study that will determine if there is a reduction in the signs and symptoms (such as back pain and stiffness) of patients with ankylosing spondylitis with infliximab therapy. This study will also study the safety of infliximab in patients with ankylosing spondylitis. The effect of infliximab on physical function, damage to joints and the quality of life in patients with ankylosing spondylitis will also be studied. Subjects received infusions of either placebo at weeks 0, 2, 6, 12, 18 and 5 mg/kg infliximab at weeks 24, 26, 30 and every 6 weeks through week 96, or 5 mg/kg infliximab at weeks 1, 2, 6, 12, 18 and every 6 weeks through week 96

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of definite Akylosing Spondylitis for at least 3 months prior to screening
* Have active disease with spinal pain
* receiving or intolerant to standard anti-inflammatory agents

Exclusion Criteria:

* Have Rheumatoid Arthritis, systemic lupus erythematosus, or other inflammatory rheumatic disease
* Have a documented history of fibromyalgia
* Have total ankylosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2002-09; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study was the proportion of subjects who achieved an ASAS 20 response at week 24.

SECONDARY OUTCOMES:
The change from baseline in BASFI at week 24, the proportion of subjects who achieved an AS major clinical response at week 24, and the change from baseline in the physical component summary score of the SF-36 at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] van der Heijde D, Han C, DeVlam K, Burmester G, van den Bosch F, Williamson P, Bala M, Han J, Braun J. Infliximab improves productivity and reduces workday loss in patients with ankylosing spondylitis: results from a randomized, placebo-controlled trial. Arthritis Rheum. 2006 Aug 15;55(4):569-74. doi: 10.1002/art.22097. PMID 16874778
- [Result] Braun J, Landewe R, Hermann KG, Han J, Yan S, Williamson P, van der Heijde D; ASSERT Study Group. Major reduction in spinal inflammation in patients with ankylosing spondylitis after treatment with infliximab: results of a multicenter, randomized, double-blind, placebo-controlled magnetic resonance imaging study. Arthritis Rheum. 2006 May;54(5):1646-52. doi: 10.1002/art.21790. PMID 16646033
- [Result] van der Heijde D, Dijkmans B, Geusens P, Sieper J, DeWoody K, Williamson P, Braun J; Ankylosing Spondylitis Study for the Evaluation of Recombinant Infliximab Therapy Study Group. Efficacy and safety of infliximab in patients with ankylosing spondylitis: results of a randomized, placebo-controlled trial (ASSERT). Arthritis Rheum. 2005 Feb;52(2):582-91. doi: 10.1002/art.20852. PMID 15692973
- [Derived] Webers C, Stolwijk C, Schiepers O, Schoonbrood T, van Tubergen A, Landewe R, van der Heijde D, Boonen A. Infliximab treatment reduces depressive symptoms in patients with ankylosing spondylitis: an ancillary study to a randomized controlled trial (ASSERT). Arthritis Res Ther. 2020 Sep 29;22(1):225. doi: 10.1186/s13075-020-02305-w. PMID 32993799
- [Derived] Braun J, Deodhar A, Dijkmans B, Geusens P, Sieper J, Williamson P, Xu W, Visvanathan S, Baker D, Goldstein N, van der Heijde D; Ankylosing Spondylitis Study for the Evaluation of Recombinant Infliximab Therapy Study Group. Efficacy and safety of infliximab in patients with ankylosing spondylitis over a two-year period. Arthritis Rheum. 2008 Sep 15;59(9):1270-8. doi: 10.1002/art.24001. PMID 18759257
- See also: A Randomized, Double-blind Trial of the Efficacy of REMICADE� (Infliximab) Compared with Placebo in Subjects with Ankylosing Spondylitis Receiving Standard Anti-inflammatory Drug Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=154&filename=CR004792_CSR.pdf
- See also: | A Randomized, Double-blind Trial of the Efficacy of REMICADE® (Infliximab) Compared with Placebo in Subjects with Ankylosing Spondylitis Receiving Standard Anti-inflammatory Drug Therap — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=154&filename=CR004792_REF1.pdf